CLINICAL TRIAL: NCT04612465
Title: Phase 3 Clinical Study to Evaluate Efficacy and Safety of ASC(Autologous Adipose-derived Stem Cells) and Fibringlue or Fibringlue in Patients With Crohn's Fistula.: A Randomized Study
Brief Title: Clinical Study to Evaluate Efficacy and Safety of ASC and Fibringlue or Fibringlue in Patients With Crohn's Fistula
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANTG-ASC-301
Record Dates: First submitted 2020-10-06; First posted 2020-11-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASC (test arm) (Experimental): (Autologous Adipose-derived Mesenchymal Stem Cells)
  Interventions: Biological: ASC
- Fibringlue (Placebo Comparator): Standard comparator
  Interventions: Drug: Fibringlue

INTERVENTIONS:
Biological: ASC — Injection of ASC(Autologous Adipose-derived Mesenchymal Stem Cells) to Crohn's Fistula.
  The ASC injection dose is about 1x10^7 cells of ASC per 1cm^2 of the surface area of the fistula, and the additional injection dose is 1.5 times the initial injection dose. and up to 30% of the ASC injection dose is administered in combination with Fibringlu.
  Other Names: (Autologous Adipose-derived Mesenchymal Stem Cells)
  Arms: ASC (test arm)
Drug: Fibringlue — Injection of Fibringlue to Crohn's Fistula. The Fibringlu injection dose is given the size of the fistula that is fill the entire fistula, and the additional injection dose is the same.
  Other Names: standard control
  Arms: Fibringlue

SUMMARY:
This is a phase III study to evaluate the efficacy and safety of ASC(Autologous Adipose-derived Stem Cells) and Fibringlue or Fibringlue in Patients With Crohn's Fistula.

DETAILED DESCRIPTION:
Experimental: ASC(Autologous Adipose-derived Stem Cells) and Fibringlue, Comparator: Fibringlue, Study type: Interventional, Study design: Randomized

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has obtained the consent of their legal representative if they are over 18 years of age and under 20 years of age.
2. Patient is diagnosed with Crohn's disease.
3. Patient who has one or more Crohn's fistulas .
4. In the case of women of childbearing potential, patient who is negative for beta-HCG pregnancy tests at the screening visit.
5. Patient is able to give written informed consent prior to study start and willing to comply with the study requirements.

Exclusion Criteria:

1. Patient who participated in other clinical trials within 30 days prior to the start of this clinical trial, or who has not passed a period equal to five times of the half-life of the drug dosed in other clinical trials.
2. Patient with a medical history or family history of Variant Creutzfeld Jakob Disease or related to this disease.
3. Patient who is sensitive to anesthetic drugs or bovine-derived materials.
4. Patient with autoimmune disease except for Crohn's disease.
5. Patient with infectious diseases such as HBV, HCV and HIV.
6. Patient with signs of Septicemia.
7. Patient with Active Tuberculosis.(Including patient with Anal Tuberculosis)
8. Pregnant or breast-feeding.
9. . Is unwilling to use an acceptable method of birth control during the whole study.
10. Patient with Inflammatory Bowel disease except for Crohn's disease.
11. Patient who is sensitive to Fibringlue.
12. Patient with a clinically relevant history of alcohol or drugs abuse, habitual smoking.
13. Patient whose adipose tissue obtained by liposuction is insufficient to manufacture the Investigational product at the intended dose.
14. Patient who is not able to understand the objective of the study or to comply with the study requirements.
15. Patient who is considered by the investigator to have a significant disease which might impact the study.
16. Patient who is considered not suitable for the study by investigator.
17. Patient who is Active Crohn's disease with CDAI 450 or higher.
18. Patient with medical history of surgery for malignant cancer in the past 5 years.(Except for carcinoma in situ)
19. Patient who exceeds 2 cm in the longest diameter of fistula.
20. Patient who dosed anti-TNF formulations such as infliximab, adalimumab, certolizumab within 3 months prior to injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who are completely blocked fistula | In the 8th week after 1st injection
  complete blockage

SECONDARY OUTCOMES:
Proportion of subjects who are completely blocked fistula | During 12 months after injection
  complete blockage
Proportion of subjects who are more than 50% blocked fistula | During 12 months after injection
  50% blockage
Score of evaluation about Investigator satisfaction using questionnaire | In the 8th week, 6th month and 12th month after final injection
  Score of evaluation about Investigator satisfaction range from 1 to 5. The lower this score, it means that the higher investigator's satisfaction with treatment effect of investigational product.
Proportion of subjects who are confirmed maintenance of fistula blockage by radiology test | Between 6th month and 12th month after final injection
  Radiology test is performed to subjects who are completely blocked fistula.
Visual improvement effect of perianal fistula wound through photography of it | Immediately before and after the injection(intervention) and during 12 months after injection(intervention)
  Visual improvement effect of perianal fistula wound is evaluated by photograph of perianal fistula wound before and after the injection(intervention).

CONTACTS AND LOCATIONS:
Overall Officials: KyuJoo Park, MD. Ph D, Principal Investigator — Seoul National University Hospital; ChangSik Yu, MD. Ph D, Principal Investigator — Asan Medical Center; YongBeom Cho, MD. Ph D, Principal Investigator — Samsung Medical Center
Locations (4):
- South Korea (4):
  - Severance, Seoul, Seodaemun-gu
  - Seoul Natinoal Univetsity Hospital, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul